CLINICAL TRIAL: NCT01128452
Title: A 4-Week, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Investigate the Safety and Efficacy of EVT 101 as Monotherapy in Patients With Treatment-Resistant Major Depression
Brief Title: Safety and Efficacy of EVT 101 in Treatment-Resistant Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Evotec has indicated that this study was discontinued due to a clinical hold issued by the FDA
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR104589; RRA-12001, EVT 101/1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: Treatment-Resistant Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- EVT 101 (Experimental): EVT 101
  Interventions: Drug: EVT 101

INTERVENTIONS:
Drug: EVT 101 — HPMC Capsule, 15 mg, once daily for 28 days
  Arms: EVT 101
Drug: Placebo — HPMC Placebo capsules, once daily for 28 days
  Arms: Placebo

SUMMARY:
This study is a 4-week, randomized, double-blind, parallel-group, placebo-controlled monotherapy study in patients with treatment-resistant major depression. After confirmation of treatment-resistance in a prospective treatment period with citalopram, each patient will be treated with either EVT 101 once daily or placebo for 28 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* Current episode of major depression that has not benefited from at least 1 but no more than 3 adequate treatment regimens
* Has as score of >/= 18 on the Ham-D-17

Exclusion Criteria:

* Pregnant or breast-feeding women
* Evidence of age-related cognitive decline or mild dementia
* At imminent risk of committing suicide
* Has with the exception of major depression, a serious medical or neurological illness, including seizure disorder, stroke, dementia, or Parkinson disease
* Has an established diagnosis of bipolar disorder, hypomania, schizoaffective disorder, major depression with psychotic features or schizophrenia
* Has had a substance or alcohol abuse or dependence disorder (except nicotine and caffeine) in the 1 year before screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Profile of EVT 101 | 28 days of EVT 101-Treatment
  AE monitoring, clinical laboratory assessments, vital sign measurements, body weight, 12-lead ECG, physical exmaninations, ophthalmological examinations and questionnaires

SECONDARY OUTCOMES:
Efficacy of EVT 101 in depression measured using the MADRS score | 28 days
  Efficacy of EVT 101 in depression measured using the MADRS score and comparing those scores at the end of treatment with scores at baseline
Percentage of patients who respond to treatment with study drug | 4 weeks
Percentage of patients who experience remission | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doris Greiling, PhD, Study Director — Evotec AG
Locations (14):
- United States (14):
  - Evotec Study Site 6, Oceanside, California
  - Evotec Study Site 19, San Diego, California
  - Evotec Study Site 15, Tampa, Florida
  - Evotec Study Site 4, Atlanta, Georgia
  - Evotec Study Site 14, Smyrna, Georgia
  - Evotec Study Site 3, Beachwood, Illinois
  - Evotec Study Site 2, Oak Brook, Illinois
  - Evotec Study Site 1, Baltimore, Maryland
  - Evotec Study Site 8, Flowood, Mississippi
  - Evotec Study Site 5, Willingboro, New Jersey
  - Evotec Study Site 9, New York, New York
  - Evotec Study Site 13, Oklahoma City, Oklahoma
  - Evotec Study Site 7, Dallas, Texas
  - Evotec Study Site 12, Houston, Texas